CLINICAL TRIAL: NCT00695331
Title: A Comparison of Titrated Oral Misoprostol Solution to Intravenous Oxytocin for Labor Augmentation: A Randomized Controlled Trial
Brief Title: Efficacy and Safety Study of Titrated Oral Misoprostol Solution for Labor Augmentation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Shi-Yann Cheng, China Medical University Beigang Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMUBH R96007; DMR96-IRB-176
Record Dates: First submitted 2008-06-08; First posted 2008-06-11 (Estimated); Last update posted 2008-07-10 (Estimated); Status verified 2008-07

CONDITIONS: Labor
Keywords: Labor Augmentation; Misoprostol; Oxytocin
MeSH Terms: interventions — Misoprostol; Oxytocin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Titrated Oral Misoprostol Solution
  Interventions: Drug: Misoprostol
- 2 (Active Comparator): Intravenous Oxytocin
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Misoprostol — Titrated Misoprostol Solution
  Other Names: Cytotec
  Arms: 1
Drug: Oxytocin — Titrated Intravenous Oxytocin
  Other Names: Piton-S
  Arms: 2

SUMMARY:
The purpose of this study is to compare the efficacy and safety of titrated oral misoprostol solution with intravenous oxytocin for labor augmentation in women without adequate uterine contractions.

DETAILED DESCRIPTION:
Numerous labor course necessitate augmentation when uterine contractions are inadequate. When the cervix is favorable, labor augmentation attempts are more likely to be successful. Augmentation is these women is traditionally undertaken with intravenous oxytocin and amniotomy, either alone or in combination.

In our previous trial, it has been proven that the method of titrated oral misoprostol is associated with a lower incidence of uterine hyperstimulation and a lower cesarean delivery rate than vaginal misoprostol for labor induction in patients with unfavorable cervix. Because administering Misoprostol solution is easy and cost saving, it is worth to develop this novel method in labor augmentation.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy between 36 and 42 weeks of gestation
* Live singleton
* Cephalic presentation
* A reassuring fetal heart rate pattern
* Bishop score greater than 6
* Inadequate uterine contraction (less than or equal to 2 per 10 minutes)

Exclusion Criteria:

* Nonreassuring fetal heart rate pattern
* Parity more than five
* Uterine scar
* Suspected placental abruption with abnormal fetal heart rate
* Vaginal bleeding other than "bloody show"
* Significant maternal cardiac, renal, or hepatic disease
* hypersensitivity to oxytocin, misoprostol or prostaglandin analogues

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 143 (Estimated)
Dates: Start 2008-02; Primary Completion 2008-12 (Estimated); Study Completion 2009-01 (Estimated)

PRIMARY OUTCOMES:
the percentage of women delivering infants vaginally within 12 hours of augmentation | post vaginal delivery

SECONDARY OUTCOMES:
uterine hyperstimulation rate | post vaginal delivery

CONTACTS AND LOCATIONS:
Overall Officials: Shi-Yann Cheng, MD, Study Chair — China Medical University Beigang Hospital
Locations (1):
- Labor Unit, Department of Obstetric and Gynecology, China Medical Univertiy Hospital, Taichung, Taiwan

REFERENCES:
- [Background] Cheng SY, Ming H, Lee JC. Titrated oral compared with vaginal misoprostol for labor induction: a randomized controlled trial. Obstet Gynecol. 2008 Jan;111(1):119-25. doi: 10.1097/01.AOG.0000297313.68644.71. PMID 18165400
- [Derived] Ho M, Cheng SY, Li TC. Titrated oral misoprostol solution compared with intravenous oxytocin for labor augmentation: a randomized controlled trial. Obstet Gynecol. 2010 Sep;116(3):612-618. doi: 10.1097/AOG.0b013e3181ed36cc. PMID 20733443
- See also: China Medical University Hospital — http://www.cmuh.org.tw